CLINICAL TRIAL: NCT01381549
Title: A Randomised, Double-blind, Dose-finding, Multicenter Study of the Safety, Tolerability, and Efficacy of GSK2251052 Therapy Compared to Imipenem-cilastatin in the Treatment of Adult Subjects With Febrile Complicated Lower Urinary Tract Infections and Acute Pyelonephritis
Brief Title: GSK2251052 in Complicated Urinary Tract Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Microbiological findings of resistance on therapy in patients with complicated urinary tract infection
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 114688
Record Dates: First submitted 2011-06-09; First posted 2011-06-27 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Infections, Urinary Tract
Keywords: Gram-negative; uropathogens; complicated lower urinary tract infection; pyelonephritis
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis | interventions — 3-(aminomethyl)-7-(3-hydroxypropoxy)-1-hydroxy-1,3-dihydro-2,1-benzoxaborole; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GSK2251052 750mg (Experimental): q12h administered via IV infusion, plus saline placebo
  Interventions: Drug: GSK2251052; Other: Placebo
- GSK2251052 1500mg (Experimental): q12h administered via IV infusion, plus saline placebo
  Interventions: Drug: GSK2251052; Other: Placebo
- imipenem-cilastatin (Active Comparator): 500 mg imipenem monohydrate and 500 mg cilastatin sodium; q6h administered via IV infusion, plus saline placebo
  Interventions: Drug: imipenem-cilastatin; Other: Placebo

INTERVENTIONS:
Drug: GSK2251052 — Reconstituted, added to 250mL 0.9% NaCl solution and administered via IV infusion
  Arms: GSK2251052 1500mg; GSK2251052 750mg
Drug: imipenem-cilastatin — Prepare as per prescribing information instructions in 100 mL bag of 0.9% NaCl and administered via IV infusion
  Other Names: Primaxin® (Manufacturer: Merck)
  Arms: imipenem-cilastatin
Other: Placebo — saline placebo

SUMMARY:
This study is being conducted to evaluate the safety, efficacy (clinical and microbiological), pharmacokinetics/pharmacodynamics of GSK2251052 and to assess whether it would be a suitable antibiotic for the treatment for febrile lower cUTI and pyelonephritis(complicated and uncomplicated). GSK2251052 will be compared to imipenem-cilastatin, which is an antibiotic commonly used to treat serious cUTI infections. GSK2251052 has a spectrum of microbiological activity that includes pathogens responsible for cUTI.

ELIGIBILITY:
Inclusion Criteria:

- Adult subjects least 18 years of age.

N.B. Females of non-childbearing or childbearing potential may be enrolled. Females of childbearing potential must have a negative pregnancy test at study entry and must have practiced adequate contraception for at least 30 days prior to study entry. Additionally, the subject agrees to one of the following methods for avoidance of pregnancy during the entire study treatment period:

* Abstinence; or,
* Oral Contraceptive, either combined estrogen/progesterone or progesterone alone, PLUS an additional barrier method [ie, condom, occlusive cap (diaphragm or cervical/vault caps) or vaginal spermicidal agent (foam/gel/film/cream/suppository)]; or,
* Injectable progesterone; or
* Implants of levonorgestrel; or,
* Estrogenic vaginal ring; or,
* Percutaneous contraceptive patches; or
* Intrauterine device (IUD) or intrauterine system (IUS) showing that failure rate is less than 1% in the IUD or IUS product label; or,
* Has a male partner who is sterilized (vasectomy with documentation of azoospermia).
* Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* Females are considered to be of non-childbearing potential if they have documented tubal ligation or hysterectomy; or are postmenopausal, defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]
* Subject requires hospitalisation and has clinical signs and symptoms of lower cUTI or pyelonephritis (complicated or uncomplicated) as defined below, that requires parenteral treatment only with a treatment course of a minimum of 5 days and a maximum of 14 days:
* Lower cUTI - subjects must have documented fever defined as >38°C oral, >38.5°C tympanic or >39°C rectal, within the last 24 hours exceptions would be:
* Afebrile subjects with lower cUTI who have a white blood cell count (WBC) ≥15,000 cells/mm3
* Afebrile subjects with a lower cUTI following requiring parenteral therapy due to a specific indication e.g. before and during an operative procedure, when oral antibiotics are not indicated or in cases where the cUTI is suspected to be due to a pathogen resistant to current oral antibiotics
* and at least two of the following UTI symptoms including dysuria, frequency, urgency or suprapubic pain, with the presence of a complicating factor:
* Male gender;
* Current bladder instrumentation or indwelling urinary catheter that has to be removed two days before the end of IV study drug administration;
* Obstructive uropathy that is expected to be medically or surgically treated during the course of IV study drug administration;
* Urogenital surgery within 7 days preceding administration of the first dose of study drug;
* Functional or anatomical abnormality of the urogenital tract including anatomic malformations or neurogenic bladder with voiding disturbance of at least 100 mL residual urine.
* Acute pyelonephritis (complicated or uncomplicated): subjects must have documented fever defined as >38°C oral, >38.5°C tympanic or >39°C rectal, within the last 24 hours and flank pain or costovertebral angle tenderness (CVA). Complicating factors for pyelonephritis are the same as for complicated UTI.
* Subject has pyuria (white blood cell [WBC] count > 10/µL (or >5/high-power field [HPF] in a conventional urinalysis) in unspun clean-catch midstream urine (MSU) or catheter urine sample or >= 10 WBC/HPF in spun MSU or catheter urine).
* Subject has Gram-negative organism(s) on direct examination of a Gram-stained specimen from unspun or spun MSU or catheter urine sample.
* Subject has provided a pre-therapy urine specimen obtained within 48 hours prior to the start of therapy, which when cultured has grown at least one and not more than two Gram-negative uropathogens at >=10^5 CFU/mL.
* A subject may be enrolled before the results of the pre-therapy urine culture is known, but the subject should be withdrawn from the study if the culture does not yield at least one but not more than two qualifying Gram-negative uropathogens at >=10^5 CFU/mL or if the culture yields Gram-positive uropathogens.
* A subject with lower cUTI or pyelonephritis (complicated or uncomplicated) who has failed a previous antibacterial treatment regimen is eligible provided a urine specimen is positive for one and not more than two bacterial Gram-negative uropathogens at >=10^5 CFU/mL. Subjects who are treatment failures due to imipenem-cilastatin should not be enrolled.
* QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block
* Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Concomitant infection requiring systemic antibacterial therapy other than study drugs at the time of randomisation.
* Subject is known to have one or more of the following:
* A urinary catheter that is not being removed during the study (or with an expectation that a catheter would be inserted during therapy with study drug and subsequently not removed during the study period; (intermittent straight catheterisation is acceptable)
* Complete permanent obstruction of the urinary tract;
* A permanent indwelling catheter or comparable instrumentation including nephrostomy that will not be removed during IV study drug administration
* Suspected or confirmed prostatitis
* Suspected or confirmed perinephric or intrarenal abscess
* A UTI suspected or confirmed to be fungal in origin (with >= 10^3 fungal CFU/mL)
* A UTI suspected or confirmed to be due to a Gram-positive uropathogen(s), with >= 10^5 Gram-positive organism CFU/mL;
* A UTI known at study entry to be caused by a pathogen(s) resistant to the study antimicrobial agent;
* Known ileal loops or vesico-ureteral reflux ;
* Polycystic kidney disease.
* Subject has an APACHE II score >20
* Subject has known severe impairment of renal function including: a calculated creatinine clearance (CrCl) of less than 50 mL/min; requirement for peritoneal dialysis, haemodialysis, or haemofiltration; oliguria (less than 20 mL urine output per hour over 24 hours);
* Subject with an intractable lower cUTI requiring more than 14 Days IV treatment.
* Subjects with asymptomatic lower cUTI, such as subjects with spinal cord injury with lower cUTI who are not able to perceive symptoms due to their injury.
* Subject with lower cUTI or pyelonephritis (complicated and uncomplicated) who has received any amount of a potentially therapeutic antibiotic within the 96 h before providing the baseline urine culture specimen or prior to the start of the study.
* Subject has Gram-positive organism(s) on direct examination of a Gram-stained specimen of spun/unspun MSU or catheter urine.
* Subject is considered unlikely to survive the 4 6 week study period or has any rapidly progressing disease or immediately life-threatening illness (including acute hepatic failure, respiratory failure or septic shock).
* Subject has evidence of known or pre-existing severe hepatic disease (Child-Pugh score of B or C).
* Subject has a known baseline haemoglobin less than 10 g/dL ,haematocrit less than 30% and/or a known reticulocyte count of >5% (i.e., reticulocytes >5% of total RBC mass)
* Subject has known neutropenia or is anticipated to develop neutropenia during the course of the study (i.e., new chemotherapy subject), with absolute neutrophil count less than 1000 cells/mm3
* Subject has a known platelet count less than 75,000 cells /mm3 (subjects with platelet counts as low as 50,000 cells /mm3 are eligible if the reduction is historically stable).
* Subject has an immunocompromising illness; including known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS), organ (including bone marrow) transplantation, hematological malignancy, and/or immunosuppressive therapy , including high-dose corticosteroids (e.g., greater than 40 mg prednisone or equivalent per day for greater than two weeks)
* Subject has participated in any investigational drug or device study within 30 days of study entry or within 5 half-lives, whichever is longer.
* Subject has previously received treatment with GSK2251052.
* Subject has a prior history of seizures or has a CNS abnormality predisposing them to seizures or has a lowered seizure threshold and/or is using concomitant medications with seizure potential.
* Subject requires probenicid or valproic acid medications.
* Subject has a history of moderate or severe hypersensitivity to beta-lactam antibiotics.
* Subject is pregnant or nursing
* Subject, in the opinion of the investigator may be significantly compromised by a potential drop in haemoglobin ≥2.5g/dl which is not related to the condition under study
* French subjects: the French subject has participated in any study using an investigational drug during the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2012-03-06 (Actual); Study Completion 2012-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- United States (4):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Corsicana, Texas
- Canada (2):
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- France (2):
  - GSK Investigational Site, Suresnes
  - GSK Investigational Site, Toulouse
- Greece (4):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Chaïdári
  - GSK Investigational Site, Goudi, Athens
  - GSK Investigational Site, Thessaloniki
- Russia (5):
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Rostov-on-Don
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, St'Petersburg
- Spain (7):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Getafe/Madrid
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Pama de Mallorca

REFERENCES:
- [Derived] O'Dwyer K, Spivak AT, Ingraham K, Min S, Holmes DJ, Jakielaszek C, Rittenhouse S, Kwan AL, Livi GP, Sathe G, Thomas E, Van Horn S, Miller LA, Twynholm M, Tomayko J, Dalessandro M, Caltabiano M, Scangarella-Oman NE, Brown JR. Bacterial resistance to leucyl-tRNA synthetase inhibitor GSK2251052 develops during treatment of complicated urinary tract infections. Antimicrob Agents Chemother. 2015 Jan;59(1):289-98. doi: 10.1128/AAC.03774-14. Epub 2014 Oct 27. PMID 25348524

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at eight centers in three countries (United States, Spain and Greece) from 28-June-2011 to 06-March-2012. A total of 20 participants were randomized in the study.
Pre-assignment Details: It was planned to enroll approximately 210 male and female participants with lower complicated urinary tract infection (cUTI) or pyelonephritis (complicated and uncomplicated); however, due to some unexpected microbiological findings, this study was terminated early with only 20 participants enrolled.
Groups:
- GSK2251052 750 mg: Eligible participants received GSK2251052, 750 milligram (mg), in 200 or 250 millilitre (mL) saline solution as intravenous (IV) infusion administered over 60 minutes, twice a day (BID) and Imipenem-cilastatin matching placebo solution, 100 mL, administered over 20 to 30 minutes, four times daily from Day 2 to Day 14 of the study.
- GSK2251052 1500 mg: Eligible participants received GSK2251052, 1500 mg, in 200 or 250 mL saline solution as IV infusion administered over 60 minutes, BID and Imipenem-cilastatin placebo solution, 100 mL, administered over 20 to 30 minutes, four times daily from Day 2 to Day 14 of the study.
- Imipenem-Cilastatin: Eligible participants received Imipenem-cilastatin 500 mg in 100 mL saline solution as IV infusion administered over 20 to 30 minutes four times daily and two doses of GSK2251052 matching placebo saline solution, 200 or 250 mL, administered over 60 minutes, BID from Day 2 to Day 14 of the study.
Period: Overall Study
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Started | 6 | 8 | 6
Completed | 6 | 8 | 5
Not Completed | 0 | 0 | 1
Not completed — Ineligible: No organisms isolated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- GSK2251052 750 mg: Eligible participants received GSK2251052, 750 mg, in 200 or 250 mL saline solution as IV infusion administered over 60 minutes, BID and Imipenem-cilastatin matching placebo solution, 100 mL, administered over 20 to 30 minutes, four times daily from Day 2 to Day 14 of the study.
- Total: Total of all reporting groups
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin | Total
Number analyzed (Participants) | 6 | 8 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (13.60) | 50.4 (24.45) | 48.0 (17.48) | 51.3 (18.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 10
  Male | 3 | 4 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 6 | 6 | 5 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters- Albumin and Total Protein
Description: Clinical laboratory parameters included albumin and total protein. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from individual post-Baseline values. Mean change from Baseline up to Late follow-up visit in albumin and total protein are presented.
Time Frame: Baseline (Day 1) to Late Follow up Visit (21 to 28 days post-IV therapy)
Population: Safety Population which comprised of all participants who received at least one dose of study medication. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram per Liter
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Gram per Liter
  Albumin: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  Albumin: On IV therapy (Day 5) | -0.5 (4.85) | -3.8 (7.09) | -0.3 (3.06)
  Albumin: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  Albumin: On IV therapy (Day 11) | 2.0 (NA) — Single participant |  |
  Albumin: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  Albumin: End of IV therapy | 1.0 (4.69) | -2.1 (7.38) | 0.8 (3.31)
  Albumin: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  Albumin: Test of Cure | 5.7 (3.67) | 1.7 (5.79) | 2.6 (2.61)
  Albumin: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  Albumin: Early Follow-up | 8.2 (2.77) | 3.5 (3.39) | 3.4 (3.65)
  Albumin: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  Albumin: Late Follow-up | 7.3 (4.93) | 3.5 (4.59) | 3.2 (3.77)
  Total protein: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  Total protein: On IV therapy (Day 5) | 0.0 (8.17) | -5.0 (9.09) | 1.0 (6.24)
  Total protein: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  Total protein: On IV therapy (Day 11) | -5.0 (NA) — Single participant |  |
  Total protein: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  Total protein: End of IV therapy | -0.4 (9.76) | -3.3 (10.14) | 3.0 (6.69)
  Total protein: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  Total protein: Test of Cure | 5.8 (7.68) | 2.1 (6.89) | 6.4 (3.29)
  Total protein: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  Total protein: Early Follow-up | 9.4 (5.13) | 5.3 (3.27) | 6.4 (4.98)
  Total protein: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  Total protein: Late Follow-up | 8.2 (4.92) | 5.3 (6.28) | 4.8 (5.40)

2. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters- Creatinine Clearance, Estimated (CCE)
Description: Clinical laboratory parameters included CCE. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from individual post-Baseline values. Mean change from Baseline up to Late follow-up visit in CCE are presented.
Time Frame: Baseline (Day 1) to Late Follow up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter per minute
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Milliliter per minute
  CCE: On IV therapy (Day 5): number analyzed (Participants) | 0 | 1 | 0
  CCE: On IV therapy (Day 5) |  | 18.0 (NA) — Single participant |
  CCE: Test of Cure: number analyzed (Participants) | 1 | 1 | 1
  CCE: Test of Cure | 2.0 (NA) — Single participant | 13.0 (NA) — Single participant | 56.0 (NA) — Single participant
  CCE: Early Follow-up: number analyzed (Participants) | 1 | 1 | 1
  CCE: Early Follow-up | 1.0 (NA) — Single participant | 21.0 (NA) — Single participant | 60.0 (NA) — Single participant
  CCE: Late Follow-up: number analyzed (Participants) | 1 | 1 | 0
  CCE: Late Follow-up | 25.0 (NA) — Single participant | 21.0 (NA) — Single participant |

3. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters- Creatinine, Direct Bilirubin and Total Bilirubin
Description: Clinical laboratory parameters included creatinine, direct bilirubin and total bilirubin. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from individual post-Baseline values. Mean change from Baseline up to Late follow-up visit in creatinine, direct bilirubin and total bilirubin are presented.
Time Frame: Baseline (Day 1) to Late Follow up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromole per liter
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Micromole per liter
  Creatinine: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  Creatinine: On IV therapy (Day 5) | -4.20 (10.347) | -5.78 (13.336) | -11.97 (10.279)
  Creatinine: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  Creatinine: On IV therapy (Day 11) | -1.50 (NA) — Single participant |  |
  Creatinine: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  Creatinine: End of IV therapy | -0.24 (13.616) | -11.26 (12.634) | -8.70 (9.426)
  Creatinine: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  Creatinine: Test of Cure | -2.17 (7.238) | -9.66 (11.743) | -8.54 (9.816)
  Creatinine: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  Creatinine: Early Follow-up | -3.90 (6.134) | 2.88 (14.662) | -4.56 (11.138)
  Creatinine: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  Creatinine: Late Follow-up | 4.43 (6.960) | -5.22 (10.760) | -5.22 (11.228)
  Total bilirubin: On IV therapy (Day 3): number analyzed (Participants) | 6 | 7 | 5
  Total bilirubin: On IV therapy (Day 3) | -7.5 (10.73) | -4.9 (4.45) | -7.2 (6.42)
  Total bilirubin: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  Total bilirubin: On IV therapy (Day 5) | -7.0 (10.18) | -3.5 (5.57) | -7.3 (8.50)
  Total bilirubin: On IV therapy (Day 8): number analyzed (Participants) | 1 | 2 | 1
  Total bilirubin: On IV therapy (Day 8) | -5.0 (NA) — Single participant | -4.5 (0.71) | -1.0 (NA) — Single participant
  Total bilirubin: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  Total bilirubin: On IV therapy (Day 11) | -1.0 (NA) — Single particpant |  |
  Total bilirubin: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  Total bilirubin: End of IV therapy | -8.2 (11.37) | -5.6 (0.71) | -5.5 (6.16)
  Total bilirubin: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  Total bilirubin: Test of Cure | -7.7 (9.14) | -4.7 (5.00) | -6.4 (7.64)
  Total bilirubin: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  Total bilirubin: Early Follow-up | -6.2 (8.29) | -4.5 (3.39) | -6.0 (7.04)
  Total bilirubin: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  Total bilirubin: Late Follow-up | -5.2 (8.73) | -4.8 (4.12) | -5.0 (4.80)

4. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters- Calcium, Carbon-dioxide (C02) Content/Bicarbonate, Chloride, Glucose, Potassium, Sodium and Urea/Blood Urea Nitrogen (BUN)
Description: Clinical laboratory parameters included C02 content/bicarbonate, chloride, glucose, potassium, sodium and urea/BUN. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from individual post-Baseline values. Mean change from Baseline up to Late follow-up visit in C02 content/bicarbonate, chloride, glucose, potassium, sodium and urea/BUN are presented.
Time Frame: Baseline (Day 1) to Late Follow up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimole per Liter
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Millimole per Liter
  Calcium: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  Calcium: On IV therapy (Day 5) | 0.082 (0.1664) | -0.112 (0.2170) | 0.060 (0.1229)
  Calcium: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  Calcium: On IV therapy (Day 11) | 0.030 (NA) — Single participant |  |
  Calcium: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  Calcium: End of IV therapy | -0.020 (0.2411) | 0.071 (0.1964) | 0.078 (0.0930)
  Calcium: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  Calcium: Test of Cure | 0.235 (0.2627) | 0.096 (0.2057) | 0.128 (0.1114)
  Calcium: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  Calcium: Early Follow-up | 0.276 (0.1383) | 0.120 (0.0919) | 0.142 (0.1232)
  Calcium: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  Calcium: Late Follow-up | 0.243 (0.0922) | 0.115 (0.1027) | 0.110 (0.1538)
  C02 content/Bicarbonate: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  C02 content/Bicarbonate: On IV therapy (Day 5) | -1.7 (3.01) | 0.0 (2.83) | -2.0 (0.00)
  C02 content/Bicarbonate: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  C02 content/Bicarbonate: On IV therapy (Day 11) | -3.0 (NA) — Single participant |  |
  C02 content/Bicarbonate: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  C02 content/Bicarbonate: End of IV therapy | -2.4 (2.07) | 0.6 (2.30) | -0.3 (2.88)
  C02 content/Bicarbonate: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  C02 content/Bicarbonate: Test of Cure | -0.8 (1.72) | 2.7 (1.80) | 1.4 (4.28)
  C02 content/Bicarbonate: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  C02 content/Bicarbonate: Early Follow-up | 0.0 (3.81) | 0.3 (1.63) | -0.4 (4.72)
  C02 content/Bicarbonate: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  C02 content/Bicarbonate: Late Follow-up | 0.7 (2.34) | 1.8 (2.71) | 1.2 (4.97)
  Chloride: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  Chloride: On IV therapy (Day 5) | 1.2 (4.07) | 1.8 (3.50) | 3.7 (1.15)
  Chloride: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  Chloride: On IV therapy (Day 11) | 4.0 (NA) — Single participant |  |
  Chloride: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  Chloride: End of IV therapy | 1.0 (3.74) | 3.0 (3.83) | -0.2 (2.32)
  Chloride: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  Chloride: Test of Cure | 0.5 (3.94) | 1.0 (3.83) | 0.2 (2.28)
  Chloride: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  Chloride: Early Follow-up | 0.6 (4.72) | 0.5 (4.51) | 0.0 (2.35)
  Chloride: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  Chloride: Late Follow-up | 0.3 (4.18) | -0.5 (3.02) | 2.2 (0.84)
  Glucose: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  Glucose: On IV therapy (Day 5) | 0.42 (1.993) | 2.25 (1.700) | -2.00 (2.685)
  Glucose: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  Glucose: On IV therapy (Day 11) | 1.50 (NA) — Single participant |  |
  Glucose: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  Glucose: End of IV therapy | -1.06 (1.372) | 1.09 (1.542) | -0.68 (2.741)
  Glucose: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  Glucose: Test of Cure | -0.35 (1.649) | -0.11 (1.173) | -0.24 (2.261)
  Glucose: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  Glucose: Early Follow-up | -0.80 (1.158) | 0.07 (1.316) | -0.78 (1.949)
  Glucose: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  Glucose: Late Follow-up | -0.45 (1.106) | 0.58 (1.703) | -0.56 (2.395)
  Potassium: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  Potassium: On IV therapy (Day 5) | 0.52 (0.662) | -0.05 (0.645) | 0.37 (0.666)
  Potassium: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  Potassium: On IV therapy (Day 11) | 0.00 (NA) — Single participant |  |
  Potassium: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  Potassium: End of IV therapy | 0.46 (0.623) | 0.24 (0.509) | 0.48 (0.407)
  Potassium: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  Potassium: Test of Cure | 0.78 (0.739) | 0.40 (0.526) | 0.44 (0.351)
  Potassium: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  Potassium: Early Follow-up | 0.40 (0.725) | 0.50 (0.400) | 0.42 (0.327)
  Potassium: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  Potassium: Late Follow-up | 0.28 (0.471) | 0.53 (0.547) | 0.40 (0.495)
  Sodium: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  Sodium: On IV therapy (Day 5) | 1.2 (2.23) | 0.3 (2.75) | 2.3 (2.52)
  Sodium: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  Sodium: On IV therapy (Day 11) | 4.0 (NA) — Single participant |  |
  Sodium: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  Sodium: End of IV therapy | 0.4 (2.79) | 1.7 (3.15) | -0.8 (2.14)
  Sodium: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  Sodium: Test of Cure | 1.8 (1.33) | 1.3 (3.40) | 1.0 (1.73)
  Sodium: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  Sodium: Early Follow-up | 1.8 (3.27) | -0.5 (3.45) | 1.0 (1.58)
  Sodium: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  Sodium: Late Follow-up | 1.2 (3.54) | -1.2 (4.36) | 2.0 (2.65)
  Urea/BUN: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  Urea/BUN: On IV therapy (Day 5) | -0.98 (2.024) | -0.45 (1.515) | -0.97 (0.874)
  Urea/BUN: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  Urea/BUN: On IV therapy (Day 11) | -2.50 (NA) — Single participant |  |
  Urea/BUN: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  Urea/BUN: End of IV therapy | -0.30 (2.633) | -1.13 (1.367) | -0.57 (1.046)
  Urea/BUN: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  Urea/BUN: Test of Cure | -0.38 (1.184) | -0.73 (1.456) | -0.38 (1.033)
  Urea/BUN: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  Urea/BUN: Early Follow-up | -0.64 (1.305) | 0.20 (2.262) | -0.34 (0.853)
  Urea/BUN: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  Urea/BUN: Late Follow-up | -0.30 (0.716) | -0.33 (1.199) | -0.12 (1.932)

5. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters- Alanine Amino Transferase (ALT), Alkaline Phosphatase (ALP), Aspartate Amino Transferase (AST), Creatine Kinase and Gamma Glutamyl Transferase (GGT)
Description: Clinical laboratory parameters included ALT, ALP, AST, Creatine kinase and GGT. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from individual post-Baseline values. Mean change from Baseline up to Late follow-up visit in ALT, ALP, AST, Creatine kinase and GGT are presented.
Time Frame: Baseline (Day 1) to Late Follow up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
International units per Liter
  ALT: On IV therapy (Day 3): number analyzed (Participants) | 6 | 7 | 5
  ALT: On IV therapy (Day 3) | 5.7 (8.14) | 10.4 (21.53) | 12.8 (11.19)
  ALT: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  ALT: On IV therapy (Day 5) | 33.2 (46.82) | 4.8 (8.85) | 13.3 (17.90)
  ALT: On IV therapy (Day 8): number analyzed (Participants) | 1 | 2 | 1
  ALT: On IV therapy (Day 8) | 4.0 (NA) — Single participant | 1.5 (6.36) | -3.0 (NA) — Single participant
  ALT: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  ALT: On IV therapy (Day 11) | 2.0 (NA) — Single participant |  |
  ALT: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  ALT: End of IV therapy | 35.4 (40.46) | 18.6 (21.35) | 21.3 (29.30)
  ALT: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  ALT: Test of Cure | 17.5 (18.53) | 7.3 (10.34) | 7.0 (10.12)
  ALT: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  ALT: Early Follow-up | 4.8 (5.97) | 1.0 (5.33) | 5.8 (7.40)
  ALT: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  ALT: Late Follow-up | 3.3 (5.99) | -0.3 (4.32) | 4.2 (5.50)
  ALP: On IV therapy (Day 3): number analyzed (Participants) | 6 | 7 | 5
  ALP: On IV therapy (Day 3) | 10.8 (26.33) | 14.3 (30.12) | 13.2 (28.28)
  ALP: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  ALP: On IV therapy (Day 5) | 11.2 (22.99) | 4.0 (27.14) | 17.7 (35.50)
  ALP: On IV therapy (Day 8): number analyzed (Participants) | 1 | 2 | 1
  ALP: On IV therapy (Day 8) | -10.0 (NA) — Single participant | 21.5 (12.02) | -10.0 (NA) — Single participant
  ALP: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  ALP: On IV therapy (Day 11) | -11.0 (NA) — Single participant |  |
  ALP: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  ALP: End of IV therapy | 7.4 (26.28) | 16.3 (34.62) | 10.2 (22.60)
  ALP: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  ALP: Test of Cure | 10.8 (23.47) | 6.9 (15.04) | 14.8 (17.01)
  ALP: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  ALP: Early Follow-up | 7.4 (21.01) | 1.2 (23.73) | 8.2 (12.01)
  ALP: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  ALP: Late Follow-up | 5.7 (20.64) | 2.3 (13.81) | 3.6 (13.13)
  AST: On IV therapy (Day 3): number analyzed (Participants) | 6 | 7 | 5
  AST: On IV therapy (Day 3) | 5.0 (12.07) | 4.1 (12.58) | 19.2 (16.04)
  AST: On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  AST: On IV therapy (Day 5) | 31.5 (57.16) | 6.3 (13.38) | 20.0 (34.66)
  AST: On IV therapy (Day 8): number analyzed (Participants) | 1 | 2 | 1
  AST: On IV therapy (Day 8) | -2.0 (NA) — Single participant | 2.0 (0.00) | 2.0 (NA) — Single participant
  AST: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  AST: On IV therapy (Day 11) | 2.0 (NA) — Single participant |  |
  AST: End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  AST: End of IV therapy | 22.0 (34.71) | 13.1 (15.08) | 15.7 (23.34)
  AST: Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  AST: Test of Cure | 1.5 (9.81) | -2.3 (4.54) | -1.4 (6.50)
  AST: Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  AST: Early Follow-up | -1.2 (8.56) | -4.8 (10.34) | 1.2 (6.76)
  AST: Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  AST: Late Follow-up | 3.3 (15.02) | -3.3 (10.07) | 3.4 (2.88)
  Creatine kinase : On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  Creatine kinase : On IV therapy (Day 5) | -76.0 (118.58) | -37.8 (46.94) | -26.0 (18.33)
  Creatine kinase : On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  Creatine kinase : On IV therapy (Day 11) | 4.0 (NA) — Single participant |  |
  Creatine kinase : End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  Creatine kinase : End of IV therapy | -36.0 (33.56) | -165.6 (407.70) | -23.7 (18.33)
  Creatine kinase : Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  Creatine kinase : Test of Cure | -65.3 (129.24) | -156.4 (420.00) | 18.4 (18.80)
  Creatine kinase : Early Follow-up: number analyzed (Participants) | 5 | 5 | 5
  Creatine kinase : Early Follow-up | -41.4 (158.04) | -218.2 (495.53) | -6.0 (30.12)
  Creatine kinase : Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  Creatine kinase : Late Follow-up | -37.8 (134.80) | -168.8 (448.90) | 0.2 (41.05)
  GGT : On IV therapy (Day 5): number analyzed (Participants) | 6 | 4 | 3
  GGT : On IV therapy (Day 5) | 41.7 (49.61) | 6.5 (8.27) | 24.0 (35.68)
  GGT : On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  GGT : On IV therapy (Day 11) | 22.0 (NA) — Single participant |  |
  GGT : End of IV therapy: number analyzed (Participants) | 5 | 7 | 6
  GGT : End of IV therapy | 35.8 (49.96) | 28.9 (39.88) | 14.0 (20.27)
  GGT : Test of Cure: number analyzed (Participants) | 6 | 7 | 5
  GGT : Test of Cure | 16.5 (20.67) | 23.3 (24.69) | 3.6 (8.76)
  GGT : Early Follow-up: number analyzed (Participants) | 5 | 6 | 5
  GGT : Early Follow-up | -1.4 (36.90) | 8.3 (13.54) | -0.8 (12.15)
  GGT : Late Follow-up: number analyzed (Participants) | 6 | 6 | 5
  GGT : Late Follow-up | -16.7 (54.70) | 1.3 (9.58) | -3.8 (12.03)

6. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to 28 days post-therapy
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Participants
  AE | 5 | 6 | 5
  SAE | 1 | 2 | 0

7. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Twelve lead ECGs were obtained during the study using an ECG machine that automatically measured PR, QRS, QT, and QT corrected by Bazett's formula (QTcB), QT corrected by Fridericia's formula (QTcF) intervals. Twelve lead ECGs were performed with the participant in a semi-supine position having rested in this position for at least 10 minutes beforehand. Measurements that deviated substantially from previous readings were repeated immediately. Three measurements were taken at pre-dose on Day 1 at least 5 min apart. One additional ECG measurement was taken after completion of the first infusion of study medication. Two ECG measurements (pre and post-1st infusion of the day) were taken on Day 4 while the participant was on IV therapy. When there was an abnormal finding, two more were taken and the mean PR interval, QRS duration, QT interval and QTcB were calculated from automated ECG readings. One ECG measurement was taken at the early safety follow-up visit.
Time Frame: Up to Late Follow-up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Participants
  Day 1: Pre-dose 1 | 0 | 4 | 2
  Day 1: Pre-dose 2 | 2 | 4 | 2
  Day 1: Pre-dose 3: number analyzed (Participants) | 5 | 7 | 6
  Day 1: Pre-dose 3 | 1 | 2 | 3
  Day 1: Post-dose | 1 | 5 | 3
  Day 4 (on IV treatment): Pre-dose: number analyzed (Participants) | 6 | 8 | 5
  Day 4 (on IV treatment): Pre-dose | 2 | 4 | 2
  Day 4 (on IV treatment): Post-dose: number analyzed (Participants) | 5 | 7 | 5
  Day 4 (on IV treatment): Post-dose | 3 | 3 | 2
  Early Follow-up: number analyzed (Participants) | 4 | 6 | 4
  Early Follow-up | 0 | 3 | 2
  Withdrawal: number analyzed (Participants) | 1 | 0 | 1
  Withdrawal | 0 | 0 | 0

8. Primary Outcome: Summary of Vital Signs: Mean Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital sign measurements included SBP and DBP (supine or semi-supine). Measurements that deviated substantially from previous readings were repeated immediately. Mean SBP and DBP are presented.
Time Frame: Up to Late Follow up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Groups:
- GSK2251052 750 mg: Eligible participants received GSK2251052, 750 mg, in 200 or 250 mL saline solution as IV infusion administered over 60 minutes, twice a day (BID) and Imipenem-cilastatin matching placebo solution, 100 mL, administered over 20 to 30 minutes, four times daily from Day 2 to Day 14 of the study.
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Millimeters of mercury (mmHg)
  SBP: Baseline (Day 1) | 129.7 (29.27) | 131.9 (14.56) | 120.0 (17.64)
  SBP: On IV therapy (Day 2) | 131.2 (15.20) | 125.4 (15.89) | 120.0 (19.75)
  SBP: On IV therapy (Day 3): number analyzed (Participants) | 6 | 8 | 5
  SBP: On IV therapy (Day 3) | 123.8 (15.09) | 126.6 (28.69) | 123.8 (13.88)
  SBP: On IV therapy (Day 4): number analyzed (Participants) | 6 | 8 | 5
  SBP: On IV therapy (Day 4) | 137.8 (17.61) | 127.0 (30.79) | 124.2 (17.98)
  SBP: On IV therapy (Day 5): number analyzed (Participants) | 6 | 7 | 5
  SBP: On IV therapy (Day 5) | 135.2 (27.58) | 126.6 (35.10) | 116.8 (18.42)
  SBP: On IV therapy (Day 6): number analyzed (Participants) | 1 | 2 | 4
  SBP: On IV therapy (Day 6) | 150.0 (NA) — Single participant | 125.5 (34.65) | 115.0 (12.25)
  SBP: On IV therapy (Day 7): number analyzed (Participants) | 1 | 2 | 3
  SBP: On IV therapy (Day 7) | 165.0 (NA) — Single participant | 125.0 (21.21) | 116.7 (20.82)
  SBP: On IV therapy (Day 8): number analyzed (Participants) | 1 | 2 | 1
  SBP: On IV therapy (Day 8) | 170.0 (NA) — Single participant | 125.0 (49.50) | 110.0 (NA) — Single participant
  SBP: On IV therapy (Day 9): number analyzed (Participants) | 1 | 1 | 1
  SBP: On IV therapy (Day 9) | 161.0 (NA) — Single participant | 130.0 (NA) — Single participant | 105.0 (NA) — Single participant
  SBP: On IV therapy (Day 10): number analyzed (Participants) | 1 | 0 | 1
  SBP: On IV therapy (Day 10) | 140.0 (NA) — Single participant |  | 110.0 (NA) — Single participant
  SBP: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  SBP: On IV therapy (Day 11) | 155.0 (NA) — Single participant |  |
  SBP: On IV therapy (Day 12): number analyzed (Participants) | 1 | 0 | 0
  SBP: On IV therapy (Day 12) | 140.0 (NA) — Single participant |  |
  SBP: On IV therapy (Day 13): number analyzed (Participants) | 1 | 0 | 0
  SBP: On IV therapy (Day 13) | 130.0 (NA) — Single participant |  |
  SBP: On IV therapy (Day 14): number analyzed (Participants) | 1 | 0 | 0
  SBP: On IV therapy (Day 14) | 152.0 (NA) — Single participant |  |
  SBP: End of IV therapy | 130.0 (17.03) | 116.1 (13.93) | 117.5 (11.73)
  SBP: Test of Cure: number analyzed (Participants) | 6 | 8 | 5
  SBP: Test of Cure | 131.3 (5.85) | 126.9 (27.17) | 126.4 (20.12)
  SBP: Early Follow-up: number analyzed (Participants) | 6 | 8 | 5
  SBP: Early Follow-up | 128.0 (17.03) | 120.1 (15.24) | 123.8 (13.10)
  SBP: Late Follow-up: number analyzed (Participants) | 6 | 8 | 5
  SBP: Late Follow-up | 148.0 (23.64) | 117.6 (21.77) | 116.6 (13.35)
  DBP: Baseline (Day 1) | 68.0 (12.84) | 77.3 (9.25) | 66.5 (4.64)
  DBP: On IV therapy (Day 2) | 78.3 (12.82) | 69.0 (15.61) | 70.3 (10.78)
  DBP: On IV therapy (Day 3): number analyzed (Participants) | 6 | 8 | 5
  DBP: On IV therapy (Day 3) | 77.2 (12.22) | 72.1 (15.72) | 71.2 (3.56)
  DBP: On IV therapy (Day 4): number analyzed (Participants) | 6 | 8 | 5
  DBP: On IV therapy (Day 4) | 85.5 (15.73) | 79.5 (19.41) | 69.6 (5.77)
  DBP: On IV therapy (Day 5): number analyzed (Participants) | 6 | 7 | 5
  DBP: On IV therapy (Day 5) | 83.8 (13.95) | 79.7 (21.89) | 67.0 (4.12)
  DBP: On IV therapy (Day 6): number analyzed (Participants) | 1 | 2 | 4
  DBP: On IV therapy (Day 6) | 90.0 (NA) — Single participant | 81.0 (12.73) | 72.5 (15.00)
  DBP: On IV therapy (Day 7): number analyzed (Participants) | 1 | 2 | 3
  DBP: On IV therapy (Day 7) | 85.0 (NA) — Single participant | 70.0 (0.00) | 67.7 (9.29)
  DBP: On IV therapy (Day 8): number analyzed (Participants) | 1 | 2 | 1
  DBP: On IV therapy (Day 8) | 90.0 (NA) — Single participant | 69.0 (15.56) | 70.0 (NA) — Single participant
  DBP: On IV therapy (Day 9): number analyzed (Participants) | 1 | 1 | 1
  DBP: On IV therapy (Day 9) | 95.0 (NA) — Single participant | 80.0 (NA) — Single participant | 65.0 (NA) — Single participant
  DBP: On IV therapy (Day 10): number analyzed (Participants) | 1 | 0 | 1
  DBP: On IV therapy (Day 10) | 69.0 (NA) — Single participant |  | 70.0 (NA) — Single participant
  DBP: On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  DBP: On IV therapy (Day 11) | 69.0 (NA) — Single participant |  |
  DBP: On IV therapy (Day 12): number analyzed (Participants) | 1 | 0 | 0
  DBP: On IV therapy (Day 12) | 75.0 (NA) — Single participant |  |
  DBP: On IV therapy (Day 13): number analyzed (Participants) | 1 | 0 | 0
  DBP: On IV therapy (Day 13) | 80.0 (NA) — Single participant |  |
  DBP: On IV therapy (Day 14): number analyzed (Participants) | 1 | 0 | 0
  DBP: On IV therapy (Day 14) | 69.0 (NA) — Single participant |  |
  DBP: End of IV therapy | 74.0 (9.94) | 69.4 (17.22) | 71.5 (12.42)
  DBP: Test of Cure: number analyzed (Participants) | 6 | 8 | 5
  DBP: Test of Cure | 82.2 (5.88) | 70.6 (12.47) | 71.8 (15.14)
  DBP: Early Follow-up: number analyzed (Participants) | 6 | 8 | 5
  DBP: Early Follow-up | 73.8 (9.62) | 72.0 (11.72) | 68.8 (12.05)
  DBP: Late Follow-up: number analyzed (Participants) | 6 | 8 | 5
  DBP: Late Follow-up | 87.7 (16.18) | 67.5 (16.13) | 65.0 (5.29)

9. Primary Outcome: Summary of Vital Signs- Mean Heart Rate
Description: Vital sign measurements included heart rate. Measurements that deviated substantially from previous readings were repeated immediately. Mean heart rate is presented.
Time Frame: Up to Late Follow-up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Beats per minute
  Baseline (Day 1) | 85.8 (10.63) | 99.3 (13.78) | 87.7 (11.78)
  On IV therapy (Day 2) | 78.2 (12.80) | 83.0 (18.97) | 81.5 (4.23)
  On IV therapy (Day 3): number analyzed (Participants) | 6 | 8 | 5
  On IV therapy (Day 3) | 77.8 (4.92) | 80.6 (14.79) | 81.4 (9.40)
  On IV therapy (Day 4): number analyzed (Participants) | 6 | 8 | 5
  On IV therapy (Day 4) | 78.5 (11.45) | 81.0 (10.43) | 73.6 (12.10)
  On IV therapy (Day 5): number analyzed (Participants) | 6 | 7 | 5
  On IV therapy (Day 5) | 72.3 (13.52) | 80.3 (10.55) | 68.2 (11.45)
  On IV therapy (Day 6): number analyzed (Participants) | 1 | 2 | 4
  On IV therapy (Day 6) | 89.0 (NA) — Single participant | 92.0 (16.97) | 74.8 (6.70)
  On IV therapy (Day 7): number analyzed (Participants) | 1 | 2 | 3
  On IV therapy (Day 7) | 81.0 (NA) — Single participant | 88.5 (16.26) | 78.3 (9.07)
  On IV therapy (Day 8): number analyzed (Participants) | 1 | 2 | 1
  On IV therapy (Day 8) | 88.0 (NA) — Single participant | 87.5 (6.36) | 82.0 (NA) — Single participant
  On IV therapy (Day 9): number analyzed (Participants) | 1 | 1 | 1
  On IV therapy (Day 9) | 84.0 (NA) — Single participant | 80.0 (NA) — Single participant | 85.0 (NA) — Single participant
  On IV therapy (Day 10): number analyzed (Participants) | 1 | 0 | 1
  On IV therapy (Day 10) | 91.0 (NA) — Single participant |  | 86.0 (NA) — Single participant
  On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  On IV therapy (Day 11) | 100.0 (NA) — Single participant |  |
  On IV therapy (Day 12): number analyzed (Participants) | 1 | 0 | 0
  On IV therapy (Day 12) | 84.0 (NA) — Single participant |  |
  On IV therapy (Day 13): number analyzed (Participants) | 1 | 0 | 0
  On IV therapy (Day 13) | 90.0 (NA) — Single participant |  |
  On IV therapy (Day 14): number analyzed (Participants) | 1 | 0 | 0
  On IV therapy (Day 14) | 92.0 (NA) — Single participant |  |
  End of IV therapy | 72.8 (11.82) | 82.8 (8.91) | 71.0 (7.32)
  Test of Cure: number analyzed (Participants) | 6 | 8 | 5
  Test of Cure | 74.5 (11.86) | 73.6 (11.94) | 74.6 (15.34)
  Early Follow-up: number analyzed (Participants) | 6 | 8 | 5
  Early Follow-up | 72.5 (11.57) | 74.0 (14.99) | 65.8 (8.90)
  Late Follow-up: number analyzed (Participants) | 6 | 8 | 5
  Late Follow-up | 76.8 (13.06) | 71.8 (11.11) | 78.2 (11.19)

10. Primary Outcome: Summary of Vital Signs- Mean Respiration Rate
Description: Vital sign measurements included respiratory rate. Measurements that deviated substantially from previous readings were repeated immediately. Mean respiration rate are presented.
Time Frame: Up to Late Follow-up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths/minute
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Breaths/minute
  Baseline (Day 1) | 17.3 (2.94) | 19.6 (3.85) | 17.3 (3.27)
  On IV therapy (Day 2): number analyzed (Participants) | 6 | 8 | 5
  On IV therapy (Day 2) | 15.0 (1.67) | 18.1 (3.68) | 16.8 (3.03)
  On IV therapy (Day 3): number analyzed (Participants) | 6 | 8 | 4
  On IV therapy (Day 3) | 14.2 (1.33) | 16.6 (3.62) | 16.8 (4.27)
  On IV therapy (Day 4): number analyzed (Participants) | 6 | 8 | 4
  On IV therapy (Day 4) | 15.5 (0.84) | 17.3 (3.99) | 17.8 (4.35)
  On IV therapy (Day 5): number analyzed (Participants) | 6 | 7 | 4
  On IV therapy (Day 5) | 14.5 (1.52) | 16.6 (3.46) | 18.8 (3.59)
  On IV therapy (Day 6): number analyzed (Participants) | 1 | 2 | 4
  On IV therapy (Day 6) | 16.0 (NA) — Single participant | 17.0 (4.24) | 16.0 (4.32)
  On IV therapy (Day 7): number analyzed (Participants) | 1 | 2 | 3
  On IV therapy (Day 7) | 16.0 (NA) — Single participant | 16.5 (3.54) | 17.3 (4.16)
  On IV therapy (Day 8): number analyzed (Participants) | 1 | 2 | 1
  On IV therapy (Day 8) | 16.0 (NA) — Single participant | 15.0 (1.41) | 20.0 (NA) — Single participant
  On IV therapy (Day 9): number analyzed (Participants) | 1 | 1 | 1
  On IV therapy (Day 9) | 14.0 (NA) — Single participant | 16.0 (NA) — Single participant | 22.0 (NA) — Single participant
  On IV therapy (Day 10): number analyzed (Participants) | 1 | 0 | 1
  On IV therapy (Day 10) | 17.0 (NA) — Single participant |  | 20.0 (NA) — Single participant
  On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  On IV therapy (Day 11) | 15.0 (NA) — Single participant |  |
  On IV therapy (Day 12): number analyzed (Participants) | 1 | 0 | 0
  On IV therapy (Day 12) | 16.0 (NA) — Single participant |  |
  On IV therapy (Day 13): number analyzed (Participants) | 1 | 0 | 0
  On IV therapy (Day 13) | 14.0 (NA) — Single participant |  |
  On IV therapy (Day 14): number analyzed (Participants) | 1 | 0 | 0
  On IV therapy (Day 14) | 14.0 (NA) — Single participant |  |
  End of IV therapy: number analyzed (Participants) | 6 | 8 | 5
  End of IV therapy | 16.0 (2.45) | 15.8 (2.96) | 16.4 (2.19)
  Test of Cure: number analyzed (Participants) | 6 | 8 | 5
  Test of Cure | 14.0 (1.79) | 15.5 (3.42) | 18.2 (4.15)
  Early Follow-up: number analyzed (Participants) | 6 | 8 | 5
  Early Follow-up | 15.3 (1.97) | 15.9 (3.52) | 16.4 (3.21)
  Late Follow-up: number analyzed (Participants) | 5 | 8 | 5
  Late Follow-up | 13.4 (1.95) | 16.0 (2.78) | 16.6 (3.71)

11. Primary Outcome: Summary of Vital Signs- Mean Temperature
Description: Vital sign measurements included temperature (oral, tympanic or rectal). Measurements that deviated substantially from previous readings were repeated immediately. Temperature was assessed as normal hospital practice dictated and the maximum daily temperature was recorded in the electronic case report form (eCRF).
Time Frame: Up to Late Follow up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Celsius
  Baseline (Day 1) | 38.08 (0.741) | 38.41 (0.946) | 38.30 (0.469)
  On IV therapy (Day 2) | 36.97 (1.063) | 37.30 (0.693) | 37.30 (0.860)
  On IV therapy (Day 3): number analyzed (Participants) | 6 | 8 | 5
  On IV therapy (Day 3) | 36.75 (0.706) | 36.79 (0.380) | 37.74 (0.817)
  On IV therapy (Day 4): number analyzed (Participants) | 6 | 8 | 5
  On IV therapy (Day 4) | 36.60 (0.469) | 36.71 (0.669) | 37.38 (0.986)
  On IV therapy (Day 5): number analyzed (Participants) | 6 | 7 | 5
  On IV therapy (Day 5) | 36.27 (0.378) | 36.59 (0.498) | 36.96 (0.654)
  On IV therapy (Day 6): number analyzed (Participants) | 1 | 2 | 4
  On IV therapy (Day 6) | 37.00 (NA) — Single participant | 36.90 (1.273) | 36.40 (0.283)
  On IV therapy (Day 7): number analyzed (Participants) | 1 | 2 | 3
  On IV therapy (Day 7) | 36.20 (NA) — Single participant | 36.95 (0.778) | 36.93 (0.416)
  On IV therapy (Day 8): number analyzed (Participants) | 1 | 2 | 1
  On IV therapy (Day 8) | 36.80 (NA) — Single participant | 36.80 (0.707) | 36.50 (NA) — Single participant
  On IV therapy (Day 9): number analyzed (Participants) | 1 | 1 | 1
  On IV therapy (Day 9) | 36.50 (NA) — Single participant | 36.80 (NA) — Single participant | 36.50 (NA) — Single participant
  On IV therapy (Day 10): number analyzed (Participants) | 1 | 0 | 1
  On IV therapy (Day 10) | 37.00 (NA) — Single participant |  | 36.50 (NA) — Single participant
  On IV therapy (Day 11): number analyzed (Participants) | 1 | 0 | 0
  On IV therapy (Day 11) | 37.00 (NA) — Single participant |  |
  On IV therapy (Day 12): number analyzed (Participants) | 1 | 0 | 0
  On IV therapy (Day 12) | 36.80 (NA) — Single participant |  |
  On IV therapy (Day 13): number analyzed (Participants) | 1 | 0 | 0
  On IV therapy (Day 13) | 36.20 (NA) — Single participant |  |
  On IV therapy (Day 14): number analyzed (Participants) | 1 | 0 | 0
  On IV therapy (Day 14) | 36.80 (NA) — Single participant |  |
  End of IV therapy | 36.18 (0.512) | 36.75 (0.676) | 36.38 (0.299)
  Test of Cure: number analyzed (Participants) | 6 | 8 | 5
  Test of Cure | 36.25 (0.418) | 35.98 (0.709) | 36.14 (0.744)
  Early Follow-up: number analyzed (Participants) | 6 | 8 | 5
  Early Follow-up | 36.23 (0.427) | 35.99 (0.387) | 36.28 (0.606)
  Late Follow-up: number analyzed (Participants) | 6 | 8 | 5
  Late Follow-up | 36.40 (0.110) | 36.08 (0.512) | 36.00 (0.394)

12. Primary Outcome: Therapeutic Response at the Test of Cure Visit
Description: The therapeutic response was the combination of a participant's clinical and microbiological response. It was assessed at the Test of Cure visit in participants who have a qualifying Gram-negative uropathogen at Baseline and have had a minimum of 5 days of IV therapy. Therapeutic response was a measure of the overall efficacy response, and a therapeutic success referred to participants who have been deemed both a 'clinical success' and a 'microbiological success'. All other combinations (other than 'clinical success' + 'microbiological success') were deemed failures for therapeutic response.
Time Frame: Test of Cure Visit (5 to 9 days post-IV therapy)
Population: Microbiological Intent to Treat (MITT) comprised of all randomized participants who received at least one dose of study medication and had at least one gram-negative uropathogen and no more than two gram-negative uropathogens (≥10^5 Colony forming units [CFU]/mL for each pathogen) identified from Baseline urine culture.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 5
Participants
  Therapeutic Success | 1 | 5 | 1
  Therapeutic Failure | 5 | 3 | 4

13. Primary Outcome: Change From Baseline in Hematology Parameters- Hematocrit
Description: Hematology parameters included hematocrit. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from individual post-Baseline values. Mean change from Baseline up to Late follow-up visit in hematocrit are presented.
Time Frame: Baseline (Day 1) to Late Follow up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Fraction
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Fraction
  End of IV therapy: number analyzed (Participants) | 5 | 8 | 6
  End of IV therapy | -0.0140 (0.06893) | -0.0155 (0.06930) | -0.0120 (0.02993)
  Late Follow-up: number analyzed (Participants) | 6 | 7 | 5
  Late Follow-up | 0.0373 (0.03079) | -0.0007 (0.03322) | -0.0038 (0.01669)

14. Primary Outcome: Change From Baseline in Hematology Parameters- Mean Corpuscle Hemoglobin (MCH)
Description: Hematology parameters included MCH. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from individual post-Baseline values. Mean change from Baseline up to Late follow-up visit in MCH are presented.
Time Frame: Baseline (Day 1) to Late Follow up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Picograms
  End of IV therapy: number analyzed (Participants) | 5 | 8 | 6
  End of IV therapy | -0.60 (0.748) | -0.60 (0.668) | -0.07 (0.628)
  Late Follow-up: number analyzed (Participants) | 6 | 7 | 5
  Late Follow-up | -0.85 (0.657) | -0.89 (0.573) | -0.14 (0.472)

15. Primary Outcome: Change From Baseline in Hematology Parameters- Mean Corpuscle Volume (MCV)
Description: Hematology parameters included MCV. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from individual post-Baseline values. Mean change from Baseline up to Late follow-up visit in MCV are presented.
Time Frame: Baseline (Day 1) to Late Follow up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Femtoliters
  End of IV therapy: number analyzed (Participants) | 5 | 8 | 6
  End of IV therapy | -3.0 (2.45) | -1.3 (1.98) | -1.0 (0.89)
  Late Follow-up: number analyzed (Participants) | 6 | 7 | 5
  Late Follow-up | -2.2 (0.98) | -1.3 (2.75) | -0.8 (1.79)

16. Primary Outcome: Change From Baseline in Hematology Parameters- Red Blood Cell (RBC) Count and Reticulocytes
Description: Hematology parameters included RBC count and reticulocytes. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from individual post-Baseline values. Mean change from Baseline up to Late follow-up visit in RBC count and reticulocytes are presented.
Time Frame: Baseline (Day 1) to Late Follow up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Trillion cells per liter
  RBC: End of IV therapy: number analyzed (Participants) | 5 | 8 | 6
  RBC: End of IV therapy | -0.10 (0.689) | -0.10 (0.707) | -0.08 (0.360)
  RBC: Late Follow-up: number analyzed (Participants) | 6 | 7 | 5
  RBC: Late Follow-up | 0.52 (0.366) | 0.07 (0.236) | 0.02 (0.228)
  Reticulocytes: End of IV therapy: number analyzed (Participants) | 5 | 8 | 6
  Reticulocytes: End of IV therapy | -0.0331 (0.04544) | -0.0312 (0.02489) | -0.0072 (0.02295)
  Reticulocytes: Late Follow-up: number analyzed (Participants) | 6 | 7 | 5
  Reticulocytes: Late Follow-up | -0.0466 (0.09881) | -0.0092 (0.03267) | 0.0080 (0.02577)

17. Primary Outcome: Change From Baseline in Hematology Parameters- Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC)
Description: Hematology parameters included hemoglobin and MCHC. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from individual post-Baseline values. Mean change from Baseline up to Late follow-up visit in hemoglobin and MCHC are presented.
Time Frame: Baseline (Day 1) to Late Follow up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram per Liter
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Gram per Liter
  Hemoglobin: End of IV therapy: number analyzed (Participants) | 5 | 8 | 6
  Hemoglobin: End of IV therapy | -3.0 (22.77) | -5.5 (21.36) | -2.5 (8.17)
  Hemoglobin: Late Follow-up: number analyzed (Participants) | 6 | 7 | 5
  Hemoglobin: Late Follow-up | 11.0 (7.24) | -2.1 (9.67) | -0.6 (4.16)
  MCHC: End of IV therapy: number analyzed (Participants) | 5 | 8 | 6
  MCHC: End of IV therapy | 4.0 (3.81) | -1.8 (6.50) | 4.2 (6.74)
  MCHC: Late Follow-up: number analyzed (Participants) | 6 | 7 | 5
  MCHC: Late Follow-up | -3.0 (8.44) | -5.0 (5.94) | 1.8 (8.29)

18. Primary Outcome: Change From Baseline in Hematology Parameters- Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet Count, Total Neutrophils and White Blood Cell Count (WBC)
Description: Hematology parameters included basophils, eosinophils, lymphocytes, monocytes, platelet count, total neutrophils and WBC. Baseline was Day 1. Change from Baseline was calculated by subtracting Baseline values from individual post-Baseline values. Mean change from Baseline up to Late follow-up visit in basophils, eosinophils, lymphocytes, monocytes, platelet count, total neutrophils and WBC are presented.
Time Frame: Baseline (Day 1) to Late Follow up Visit (21 to 28 days post-IV therapy)
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gigacells per Liter
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 6
Gigacells per Liter
  Basophils: End of IV therapy: number analyzed (Participants) | 5 | 8 | 5
  Basophils: End of IV therapy | 0.028 (0.0084) | 0.018 (0.0116) | 0.014 (0.0182)
  Basophils: Late Follow-up: number analyzed (Participants) | 6 | 7 | 5
  Basophils: Late Follow-up | 0.022 (0.0147) | 0.020 (0.0163) | 0.016 (0.0114)
  Eosinophils: End of IV therapy: number analyzed (Participants) | 5 | 8 | 5
  Eosinophils: End of IV therapy | 0.274 (0.1389) | 0.096 (0.0980) | 0.090 (0.0682)
  Eosinophils: Late Follow-up: number analyzed (Participants) | 6 | 7 | 5
  Eosinophils: Late Follow-up | 0.093 (0.1488) | 0.067 (0.0966) | 0.086 (0.0385)
  Lymphocytes: End of IV therapy: number analyzed (Participants) | 5 | 8 | 5
  Lymphocytes: End of IV therapy | 0.580 (1.2076) | 0.514 (0.3816) | 0.596 (0.5140)
  Lymphocytes: Late Follow-up: number analyzed (Participants) | 6 | 7 | 5
  Lymphocytes: Late Follow-up | 0.687 (1.5191) | 0.774 (0.4808) | 0.436 (0.7578)
  Monocytes: End of IV therapy: number analyzed (Participants) | 5 | 8 | 5
  Monocytes: End of IV therapy | -0.188 (0.3739) | -0.256 (0.2015) | -0.442 (0.3841)
  Monocytes: Late Follow-up: number analyzed (Participants) | 6 | 7 | 5
  Monocytes: Late Follow-up | -0.380 (0.4553) | -0.230 (0.3902) | -0.186 (0.2103)
  Platelet count: End of IV therapy: number analyzed (Participants) | 5 | 6 | 5
  Platelet count: End of IV therapy | 141.0 (171.58) | 83.2 (139.06) | 105.4 (92.20)
  Platelet count: Late Follow-up: number analyzed (Participants) | 6 | 5 | 5
  Platelet count: Late Follow-up | 48.8 (129.10) | 45.4 (34.93) | 39.8 (35.81)
  Total neutrophils: End of IV therapy: number analyzed (Participants) | 5 | 8 | 5
  Total neutrophils: End of IV therapy | -8.178 (3.6642) | -6.695 (4.6214) | -4.656 (6.6652)
  Total neutrophils: Late Follow-up: number analyzed (Participants) | 6 | 8 | 5
  Total neutrophils: Late Follow-up | -6.765 (4.0488) | -7.737 (6.3494) | -7.902 (8.1795)
  WBC count: End of IV therapy: number analyzed (Participants) | 5 | 8 | 5
  WBC count: End of IV therapy | -7.48 (4.242) | -6.30 (4.607) | -4.36 (6.696)
  WBC count: Late Follow-up: number analyzed (Participants) | 6 | 7 | 5
  WBC count: Late Follow-up | -6.33 (4.918) | -7.11 (6.207) | -7.54 (8.486)

19. Secondary Outcome: Microbiological Response at the End of IV Therapy Visit, Test of Cure Visit and Late Follow-Up Visit
Description: Microbiological response involved both microbiological success and microbiological failure. A reduction in the uropathogens in the urine culture and no growth on blood culture was termed as microbiological success. Increase in the uropathogens in the urine culture and pathogens identified in the blood culture or use of antibacterials other than study treatments were classified as microbiological failures.
Time Frame: End of IV therapy (0-24 hours post-therapy), Test of Cure Visit (5 to 9 days post-IV therapy) and Late Follow-up (21-28 days post-therapy)
Population: MITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 5
Participants
  End of IV therapy: Microbiological Success | 3 | 5 | 5
  End of IV therapy: Microbiological Failure | 3 | 3 | 0
  Test of Cure: Microbiological Success | 1 | 5 | 1
  Test of Cure: Microbiological Failure | 5 | 3 | 4
  Late Folllow-up: Microbiological Success | 2 | 6 | 1
  Late Folllow-up: Microbiological Failure | 4 | 2 | 4

20. Secondary Outcome: Clinical Response at the End of IV Therapy Visit, Test of Cure Visit and Late Follow-Up Visit
Description: Clinical response was a combination of clinical success and clinical failure. In clinical success, participants showed no signs and symptoms of pyelonephritis and lower complicated urinary tract infection and antibiotics are not used for the same. In clinical failure, there is reappearance of signs and symptoms of and lower complicated urinary tract infection and participant required antibiotics for the same.
Time Frame: as for outcome 19
Population: MITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 5
Participants
  End of IV therapy: Clinical Success | 4 | 6 | 5
  End of IV therapy: Clinical Failure | 2 | 2 | 0
  Test of Cure: Clinical Success | 4 | 6 | 4
  Test of Cure: Clinical Failure | 2 | 2 | 1
  Late Follow-up: Clinical Success | 3 | 6 | 2
  Late Follow-up: Clinical Failure | 3 | 2 | 3

21. Secondary Outcome: Therapeutic Response (Combined Clinical and Microbiological Response) at the End of IV Visit and Late Follow-Up Visit
Description: as for outcome 12
Time Frame: End of IV therapy (0-24 hours post-therapy) and Late Follow-up (21-28 days post-therapy)
Population: MITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 6 | 8 | 5
Participants
  End of IV therapy: Therapeutic Success | 3 | 5 | 5
  End of IV therapy: Therapeutic Failure | 3 | 3 | 0
  Late Follow-up: Therapeutic Success | 2 | 6 | 1
  Late Follow-up: Therapeutic Failure | 4 | 2 | 4

22. Secondary Outcome: Maximum Plasma Concentration (Cmax) of GSK2251052
Description: The planned pharmacokinetic (PK) and PK/pharmacodynamic analyses were not performed, because the PK data was not collected.
Time Frame: Day 3: Pre- dose (just prior to the start of the first infusion of the day) and 1 hour (just prior to the end of the infusion), 2, 4, and 12 hours post-dose
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Area Under the Concentration Time Curve (AUC) of GSK2251052
Description: as for outcome 22
Time Frame: as for outcome 22
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Time to Cmax (Tmax) of GSK2251052
Description: as for outcome 22
Time Frame: as for outcome 22
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Cmax of GSK2251052 Using Non-intensive PK Sampling
Description: as for outcome 22
Time Frame: Day 4: Pre- dose (just prior to the start of the first infusion of the day) and 1 hour (just prior to the end of the infusion), 2, 4, and 12 hours post-dose
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 0 | 0 | 0

26. Secondary Outcome: AUC of GSK2251052 Using Non-intensive PK Sampling
Description: as for outcome 22
Time Frame: as for outcome 25
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 0 | 0 | 0

27. Secondary Outcome: Tmax of GSK2251052 Using Non-intensive PK Sampling
Description: as for outcome 22
Time Frame: as for outcome 25
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 0 | 0 | 0

28. Secondary Outcome: Cmax of GSK2251052 Using Intensive PK Sampling
Description: as for outcome 22
Time Frame: Day 4: Pre-dose (just prior to the start of the first infusion of the day) 0.5, 1 hour (just prior to the end of the infusion), 1.25, 1.5, 2, 3, 4, 8 and 12 hours post-dose
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 0 | 0 | 0

29. Secondary Outcome: AUC of GSK2251052 Using Intensive PK Sampling
Description: as for outcome 22
Time Frame: as for outcome 28
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 0 | 0 | 0

30. Secondary Outcome: Tmax of GSK2251052 Using Intensive PK Sampling
Description: as for outcome 22
Time Frame: as for outcome 28
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 days post-therapy
Description: SAE and non-SAE are reported for the Safety population which consisted of all participants who received at least one dose of study medication.
Arm/Group | GSK2251052 750 mg | GSK2251052 1500 mg | Imipenem-Cilastatin
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/8 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 5/8 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2251052 750 mg (N=6) | GSK2251052 1500 mg (N=8) | Imipenem-Cilastatin (N=6)
Aspiration bronchial (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2251052 750 mg (N=6) | GSK2251052 1500 mg (N=8) | Imipenem-Cilastatin (N=6)
Nausea (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Papillitis (General disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.